CLINICAL TRIAL: NCT07245394
Title: SHIFT-IBD: Switching to High-efficacy Anti-IL-23 Guselkumab in Ustekinumab-exposed Persons With Active IBD
Brief Title: Switching to the IL-23 Inhibitor Guselkumab for People With Active IBD Who Previously Used Ustekinumab (SHIFT-IBD)
Acronym: SHIFT-IBD
Status: Recruiting | Type: Observational
Sponsor: TIDHI Innovation Inc. (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TIDHI_001; ISRCTN13202059 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2025-09-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn Disease (CD); Ulcerative Colitis (UC); IBD-unclassified (IBD-U)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — guselkumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Early Switch Cohort (ESC): Patients with CD or UC who had inadequate response to on-label maintenance ustekinumab (90 mg every 8 weeks) that requires a change in advanced therapy, as determined by the treating physician. Inadequate response could be either loss of response, partial response, or persistent endoscopic activity.
  Interventions: Biological: Guselkumab (Tremfya)
- Exhausted Ustekinumab Cohort (EUC): Patients with CD or UC who had inadequate response to off-label maintenance ustekinumab (90 mg every 6 or 4 weeks) that requires a change in advanced therapy, as determined by the treating physician. Inadequate response could be either loss of response, partial response, or persistent endoscopic activity.
  Interventions: Biological: Guselkumab (Tremfya)

INTERVENTIONS:
Biological: Guselkumab (Tremfya) — Switching to Guselkumab (Tremfya) in People With Active IBD Previously Treated With Ustekinumab.

SUMMARY:
The SHIFT-IBD Study is being conducted at multiple medical centers across Canada to evaluate how well guselkumab (Tremfya) works for people with inflammatory bowel disease (IBD) who haven't responded well enough to ustekinumab.

Patients will begin guselkumab based on their doctor's decision. If eligible, they may be invited to participate in the study, which involves monitoring symptoms, test results, and overall health over the course of one year.

Guselkumab will be given according to local medical guidelines. Doctors can adjust the treatment as needed, just like in routine care.

Researchers believe that switching to guselkumab may be as effective as other advanced treatments. For those who saw some improvement on ustekinumab but not enough, guselkumab may offer better symptom control-without worsening results on medical tests like endoscopy.

The goal is to explore better treatment options for people whose IBD has not been well controlled with current therapies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any gender aged ≥ 18.
* Confirmed diagnosis of IBD (CD, UC, or IBDU) for at least 6 months prior to baseline visit. Subjects with IBDU will be grouped with subjects with UC. The CD proportion of patients will be capped at 75%.
* Subjects have received ustekinumab for at least 14 weeks and who are currently on or recently discontinued ustekinumab therapy.
* For subjects that have recently discontinued ustekinumab, the last dose of ustekinumab must have been within 12 weeks before Week 0, and no other advanced therapy (i.e., infliximab, adalimumab, golimumab, certolizumab pegol, vedolizumab, natalizumab, risankizumab, mirikizumab, tofacitinib, upadacitinib, ozanimod, etrasimod) was started since stopping ustekinumab.
* Subjects with an inadequate response to ustekinumab who require a change in advanced therapy and are initiating guselkumab, as determined by the treating physician.
* For subjects on off-label ustekinumab dosing (90 mg every 4 or 6 weeks (off-label dosing), enrollment will be capped at 60%.
* Ability and willingness to give written informed consent and comply with the requirements of this study protocol.
* Subjects who have evidence of ongoing endoscopic evidence of disease activity within 3 months prior to Week 0, defined as:

  * For Crohn's Disease: Colonoscopy showing SES-CD score (excluding the presence of narrowing component) of ≥6 (or ≥4 for participants with isolated ileal disease), OR presence of ulcers larger than 5 mm in any segment.
  * For Ulcerative Colitis: Colonoscopy showing Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score ≥4, OR presence of erosions or ulcers in any segment.

Exclusion Criteria:

* History of prior exposure to any anti-p19 inhibitor (risankizumab or mirikizumab).
* Subjects with formal contraindication to guselkumab per the drug label.
* Use of guselkumab for an off-label indication, dosing regimen, or route of administration. Subjects who did not receive guselkumab induction will be excluded.
* Subjects with an ostomy or ileo-anal pouch.
* Subjects with a history of bowel surgery within 6 months prior to Week 0.
* Subjects displaying clinical signs of acute severe UC, fulminant colitis or toxic megacolon within 3 months prior to Week 0.
* Subjects who are expected to require bowel surgery by their IBD physician within the year of enrollment.
* Subjects on 1 or more concomitant biologics.
* Subjects with a history of colonic dysplasia (low-grade dysplasia, high-grade dysplasia, or colorectal cancer). Note: Patients with a history of indefinite for dysplasia would be eligible.
* Subjects with formal contraindication or unwilling to undergo lower endoscopy.
* The patient is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients who had inadequate response to ustekinumab and switched therapy to guselkumab.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of participants achieving deep remission in IBD patients treated with guselkumab after switching from ustekinumab | Week 52
  Deep remission is defined as both absence of symptomatic worsening and endoscopic remission.
  Outcomes will be reported as the proportion of participants achieving deep remission at Week 52.
Rate of participants achieving deep remission, stratified by cohorts | Week 52
  Deep remission is defined as both absence of symptomatic worsening and endoscopic remission.
  Outcomes will be reported as the proportion of participants achieving deep remission at Week 52 and stratified by Early Switch Cohort (ESC) and Exhausted Ustekinumab Cohort (EUC).

SECONDARY OUTCOMES:
Rate of participants with absence of symptomatic worsening | Week 52
  Absence of symptomatic worsening defined as the absence of:
  1. For Crohn's disease: An increase of 30 percent or more in the average daily stool frequency score (SFS) and/or an increase of 30 percent or more in the average daily abdominal pain score (APS) compared to Baseline.
  2. For ulcerative colitis: An increase of 30 percent or more in the average daily stool frequency score (SFS) and/or an increase of 30 percent or more in the average daily rectal bleeding score (RBS) compared to Baseline.
Rate of participants achieving endoscopic remission | Week 52
  Endoscopic remission is defined as follows:
  1. For Crohn's disease: A Simple Endoscopic Score for Crohn's Disease (SDS-CD) of 4 or less, or a score of 2 or less in the ileal segment (excluding the narrowing component) in cases of disease limited to the ileum, with an ulceration subscore of 0.
  2. For ulcerative colitis: A Ulcerative Colitis Endoscopic Index of Severity (UCEIS) of 1 or less, with a bleeding subscore of 0 and an erosions/ulcers subscore of 0.
Rate of participants achieving endoscopic response | Week 52
  Endoscopic response is defined as follows:
  1. For Crohn's disease: A reduction of 50 percent or more in the Simple Endoscopic Score for Crohn's Disease (SDS-CD) compared to Baseline (excluding the narrowing component).
  2. For ulcerative colitis: A reduction of 2 points or more in the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) compared to baseline.
Rate of participants with absence of symptomatic worsening | Any study visit (Week 4, Week 12, Week 32, Week 52)
  Absence of symptomatic worsening defined as the absence of:
  1. For Crohn's disease: An increase of 30 percent or more in the average daily stool frequency score (SFS) and/or an increase of 30 percent or more in the average daily abdominal pain score (APS) compared to the baseline value.
  2. For ulcerative colitis: An increase of 30 percent or more in the average daily stool frequency score (SFS) and/or an increase of 30 percent or more in the average daily rectal bleeding score (RBS) compared to Baseline.
Rate of participants achieving symptomatic remission among those not in remission at baseline | Week 12 and Week 52
Rate of participants achieving steroid-free remission among corticosteroid users at baseline | Week 52
  Steroid-free remission defined as no corticosteroid use and meeting symptomatic remission criteria
Rate of participants discontinuing guselkumab therapy | Any study visit (Week 4, Week 12, Week 32, Week 52)

OTHER OUTCOMES:
Rate of participants achieving early symptomatic response among those not in symptomatic remission at baseline | Week 4
  Early symptomatic response at week 4 among patients who were not in symptomatic remission at baseline is defined as follows:
  1. For Crohn's disease: A decrease of 30 percent or more in the average daily stool frequency score (SFS) and/or a decrease of 30 percent or more in the average daily abdominal pain score (APS), with both scores not worse than Baseline.
  2. For ulcerative colitis: An increase of 30 percent or more in the average daily stool frequency score (SFS) and/or an increase of 30 percent or more in the average daily rectal bleeding score (RBS) compared to Baseline.
Rate of participants achieving biochemical remission | Week 52
  Biochemical remission at among patients with available fecal calprotectin (FCAL) and C-reactive protein (CRP).
  Biochemical remission is defined as FCAL ≤250 ug/g AND a CRP ≤5 mg/L among patients with available either an elevated FCAL or CRP at baseline.
Rate of participants achieving biochemical remission | Week 12
  Biochemical remission at among patients with available fecal calprotectin (FCAL) and C-reactive protein (CRP).
  Biochemical remission is defined as FCAL ≤250 ug/g AND a CRP ≤5 mg/L among patients with available either an elevated FCAL or CRP at baseline.
Change from baseline in quality of life | Week 52
  Quality of Life (QoL) outcomes will be reported as the change from baseline, using the following assessments:
  EuroQoL 5-Dimension 5-Level questionnaire (EQ-5D-5L): This tool evaluates five dimensions of health, each rated on a scale from 1 to 5. Higher scores indicate worse health status.
  Short Form Health Survey (SF-36): This questionnaire measures eight health domains, with each domain scored from 0 to 100. Higher scores reflect better health status.
Change from baseline in work productivity | Week 52
  Work Productivity outcomes will be reported as the change from baseline, assessed using the Work Productivity and Activity Impairment questionnaires specific to Crohn's disease (WPAI-CD) and ulcerative colitis (WPAI-UC). Scores range from 0 to 100 percent, with higher percentages indicating greater impairment in work and daily activities.
Change from baseline in mental health (anxiety) | Week 52
  Mental Health (anxiety) outcomes will be reported as the change from baseline, assessed using the Generalized Anxiety Disorder 7-item Scale (GAD-7): Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change from baseline in mental health (depression) | Week 52
  Mental Health (depression) outcomes will be reported as the change from baseline, assessed using the Patient Health Questionnaire-9 (PHQ-9): Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Change from baseline in fatigue | Week 52
  Fatigue outcomes will be reported as the change from baseline, assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue scale (FACIT-F). Scores range from 0 to 52, with higher scores indicating less fatigue and better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Laura E. Targownik, MD, MSHS, FRCPC, Principal Investigator — TIDHI Innovation Inc.; Mark Silverberg, MD, PhD, FRCPC, Principal Investigator — TIDHI Innovation Inc.
Locations (9):
- Canada (9):
  - MA MacMillan, Fredericton, New Brunswick
  - Barrie GI Associates, Barrie, Ontario
  - Brampton Gastroenterology Research Group Inc, Brampton, Ontario
  - GNRR Digestive Clinics and Research Center Inc., Brampton, Ontario
  - LDDI Clinical Trials Inc. dba London Digestive Disease Institute, London, Ontario
  - West Gta Research Inc., Mississauga, Ontario
  - Abp Research Services Corporation, Oakville, Ontario
  - Taunton Surgical Center, Oshawa, Ontario
  - Toronto Immune and Digestive Health Institute, Toronto, Ontario